CLINICAL TRIAL: NCT06185114
Title: Periodontal Inflammation and Wound Healing in Multiple Extractions
Status: Withdrawn | Type: Observational
Why Stopped: Study no longer focus of laboratory/group of researchers
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0886-23-EP
Record Dates: First submitted 2023-12-11; First posted 2023-12-29 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Wound Heal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples will be taken and retained for either scRNA sequencing and/or flow cytometry.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Young (ages 21-50) requiring multiple extractions: Participants aged 21-50 requiring multiple extractions will be consented. These participants will undergo soft tissue, gingival crevicular fluid (GCF), venous blood sampling and cone beam commuted tomography (CBCT) analysis to determine age-related factors associated with post-extraction wound healing.
- Old (ages 65-80) requiring multiple extractions: Participants aged 65-80 requiring multiple extractions will be consented. The older participants will undergo soft tissue, gingival crevicular fluid (GCF), venous blood sampling and cone beam commuted tomography (CBCT) analysis to determine age-related factors associated with post-extraction wound healing.

SUMMARY:
Four participants requiring multiple dental extractions will be recruited for this study. Two participants will be 21-50 years old, two participants will be 65-80 years old. Following tooth extractions, soft tissue sampling will be completed from the extraction sockets at baseline, one week, two weeks and three weeks post-extraction. Soft tissue will be processed for sc-RNA sequencing and/or flow cytometry to determine what cells, genomic pathways are present at various timepoints during wound healing following dental extractions.

DETAILED DESCRIPTION:
The purpose of this study is to better understand the cellular and immunological events occurring at various time points following dental tooth extractions as it relates to age of participants. Four participants requiring multiple extractions prior to denture fabrication will be enrolled: two will be younger than 50 years old, two will be older than 65. Inclusion criteria include: participants seeking multiple tooth extractions due to advanced bone loss or non-restorable teeth. Prior to tooth extraction, baseline clinical and radiographic data will be collected; including participant's height and weight, gingival crevicular fluid sampling (GCF), HbA1c reading, saliva sampling peripheral blood draw and smoking status. Routine, atraumatic extraction of the teeth under local anesthetic will be performed. Following extraction, a 3 mm x 3 mm soft tissue sample will be collected from one of the extraction sites and frozen/processed for sc-RNA sequencing and/or flow cytometry; the extraction sites will be sutured closed. The participants will return to clinic in one week's time for suture removal and soft tissue sampling of an adjacent previously unsampled extraction site under local anesthetic. The participants will return to clinic in another week's time (two weeks post-extraction) for a third soft tissue sample under local anesthetic from a previously unsampled extraction site. All soft tissue samples will be processed for scRNA sequencing and or flow cytometry. At all soft tissue sampling appointments, wound fluid will be collected from the extraction sites and processed for biomarkers via multiplex. Saliva samples will be frozen at time of sampling and will be frozen for multiplex evaluation. The single blood draw will be processes via sc-RNA sequencing and/or flow cytometry to assess presence of systemic immune cells. Final evaluation will be 3 months post-extraction and will include clinical (PD, BOP, CAL) and radiographic (CBCT) data collection. Statistical analyses will be completed to determine associations between various time points in the wound healing process and variables of interest (age, gender, etc), clinical measures, including body mass index (BMI) and outcomes (endotypes, measures of healing).

ELIGIBILITY:
Inclusion Criteria:

* requires multiple dental extractions
* aged 21-50, 65-80 years old

Exclusion Criteria:

* history of systemic inflammatory diseases or medications

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Four participants seeking multiple dental extractions; 21-50 years old, 65-80 years old.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Inflammatory Cells | Baseline, 1 week, 2 weeks, 3 weeks
  Presence or absence of inflammatory cells

CONTACTS AND LOCATIONS:
Overall Officials: Amy C Killeen, DDS, MS, Principal Investigator — University of Nebraska

IPD SHARING:
Plan to Share IPD: No